CLINICAL TRIAL: NCT05588752
Title: Efficacy of Transverse Abdominal Plane Block (TAP Block) With Bupivacaine and Dexamethasone for the Management of Post-cesarean Pain at the CHU Sourô Sanou (CHUSS) in Bobo-Dioulasso
Brief Title: Transverse Abdominal Plane Block for Caesarean
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université NAZI BONI (Other)
Responsible Party: Principal Investigator, Ismael Guibla, Clinical doctor, Université NAZI BONI
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: INSSA 2
Record Dates: First submitted 2022-10-16; First posted 2022-10-20 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Caesarean Section; Pain
Keywords: Caesarean, TAP-block, Postoperative pain
MeSH Terms: conditions — Pain; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Patients admitted for caesarean under spinal anesthesia were randomized according to the sealed envelope method into two groups. Group 1 received 100 µg of morphine intrathecally at induction and group 2 a bilateral TAP block at the end of cesarean section with 20 ml of bupivacaine 0.25% and dexamethasone 4 mg in the same syringe on each side.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (No Intervention): will receive at induction of spinal anesthesia 100 µg of morphine
- group 2 (Experimental): No morphine in spinal anesthesia but will receive a bilateral TAP block with 20 ml of Bupivacaine 0.25% and dexamethasone 4 mg in the same syringe on each side
  Interventions: Other: TAP block

INTERVENTIONS:
Other: TAP block — TAP block under ultrasound
  Arms: group 2

SUMMARY:
Cesarean sectionis a commonly performed major surgical procedure that results in significant postoperative pain. The objective of this study was to evaluate the effectiveness in the management of post-cesarean pain at the CHU Souro Sanou of Bobo-Dioulasso

ELIGIBILITY:
Inclusion Criteria:

* Adult parturients (≥ 18 years old) awaiting caesarean section under spinal anesthesia
* ASAI, ASAII

Exclusion Criteria:

* Lack of informed consent,
* Parturients with cognitive disorders,
* Parturients with notion of chronic pain,
* Allergy to local anesthetics,
* Morphine allergy
* Parturients not understanding pain assessment scores

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Proportion of mild pain on mobilization in the first 24 postoperative hours | Hours 24 postoperative
  The numerical pain score after moving from a lying position to a sitting position

SECONDARY OUTCOMES:
Proportion of mild pain at rest in the first 24 postoperative hours | Hours 24 postoperative
  The numerical pain score at rest
Proportion of mild pain on mobilization in the first 48 postoperative hours | Hours 48 postoperative
  The numerical pain score after moving from a lying position to a sitting position
Proportion of nausea-vomiting postoperative during the first 48 hours | Hours 48 postoperative
  At each passage of the nurses
Proportion of maternal satisfaction during the first 48 hours postoperatively | Hours 48 postoperative
  The simple numerical score

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Souro Sanou, Bobo-Dioulasso, Houet, Burkina Faso

IPD SHARING:
Plan to Share IPD: No